CLINICAL TRIAL: NCT02812550
Title: Impact of Full-spectrum Endoscopy in Colorectal Cancer Screening: Randomized Controlled Trial
Brief Title: Full-spectrum Endoscopy in Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Mª Henar Núñez Rodriguez, Dra Mª Henar Núñez Rodriguez, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: GRS 1073/A/15
Record Dates: First submitted 2016-06-15; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
Keywords: full-spectrum endoscopy; polyp detection rate; colorectal cancer; colorectal screening; adenoma detection rate; endoscopic innovations
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- full-spectrum colonoscopy (Other): Colonoscopy is performed with a full-spectrum colonoscopy (330º angle of view)
  Interventions: Procedure: colonoscopy procedure
- standar forward-viewing colonoscopy (Other): Colonoscopy is performed with standar forward-viewing colonoscopy (170º angle of view)
  Interventions: Procedure: colonoscopy procedure

INTERVENTIONS:
Procedure: colonoscopy procedure — endoscopy performed with a standard forward view colonoscopy or with full-spectrum endoscopy

SUMMARY:
The purpose of this study is to compare the adenoma detection rates of full-spectrum endoscopy versus standard forward-viewing colonoscopy in colorectal cancer screening programme.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common neoplasia and the second leading cause of cancer death in West countries. Colonoscopy is the gold standard for prevention of colorectal cancer disease. Screening for colorectal cancer with biennial faecal occult blood testing is a widely used strategy followed by colonoscopy for those with a positive test. Colonoscopy identifies polyps during the procedure as well as polyp removal in order to prevent progression to cancer. Although, interval cancer appears after a colonoscopy because of 22-28% of polyp missed rates. Advanced Technology may improve adenoma detection rates so decrease interval cancer and reduce mortally. Full-spectrum endoscopy with 330º angle vision decrease adenoma miss rate in general population.

The investigators conducted a randomized trial in patients from colorectal cancer screening programme (aged 50-69 years) after faecal immunological test positive. One arm the colonoscopy is performed with standard forward view colonoscopy (170º angle view) and the other arm is performed with full-spectrum endoscopy (EndoChoice) (330º angle view)

ELIGIBILITY:
Inclusion Criteria:

* patient referred for colorectal cancer screening with positive fecal inmunological test.
* Age between 50 and 69 years

Exclusion Criteria:

* history of colonic resection,
* high risk for colorectal cancer like family history of colorectal cancer o polyposis syndrome,
* inflammatory bowel disease,
* patients with lower gastrointestinal bleeding symptoms,
* acute diverticulitis,
* colonic strictures,
* poor bowel preparation (Boston scale less than 5 points)

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate in the two different colonoscopies | one week
  number of colonoscopies at wich one or more histologically confirmed adenomas were found divided by the total number of colonoscopies performed in the same time period.

SECONDARY OUTCOMES:
time to caecal intubation in each group | one week
  time to reach appendicular orifice
total procedure time in each group | one week
  time since the begining of the procedure till is totally finish
Adverse events | one week
  Any inmediatly complication
advance adenoma rate in each group | one week
  10mm or greater in size, villous component or high grade dysplasia
polyp detection rate in right and left colon in each group | one week
polyp retrieval rate in each group | one week
  proportion of resected polyps that were retrieved and sent for histologically analysis
caecal intubation rate in each group | one week
  proportion of all colonoscopic procedures in which the caecum, terminal ileum was reached
colonoscopy withdrawal time | one week
  average time taken withdraw the colonoscope from the caecal pole to the anus.

CONTACTS AND LOCATIONS:
Overall Officials: Mª Henar Núñez Rodriguez, MD, PhD, Principal Investigator — Hospital del Rio Hortega Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nunez-Rodriguez H, Diez-Redondo P, Perez-Miranda M, Gonzalez Sagrado M, Conde R, De la Serna C. Role of Full-spectrum Endoscopy in Colorectal Cancer Screening: Randomized Trial. J Clin Gastroenterol. 2019 Mar;53(3):191-196. doi: 10.1097/MCG.0000000000000975. PMID 29283904